CLINICAL TRIAL: NCT00749697
Title: Investigating Absorbed Radiation Dose Delivered to Differentiated Thyroid Cancer Metastases Following Administration of Fixed Activity of Radioactive Iodine
Brief Title: Radioiodine Dosimetry Protocol for Thyroid Cancer Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Dr Kate Newbold, Royal Marsden NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CCR3047
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2008-09-09 (Estimated); Status verified 2008-09

CONDITIONS: Thyroid Carcinoma; Metastatic Sites Lung Bone Nodal
Keywords: radioiodine; differentiated thyroid cancers; dosimetry; metastases
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: SPECT scan — SPECT scan measures the amount of radio activity that is remaining in patients' body after the consumption of radio iodine for therapeutic purpose

SUMMARY:
The main purpose of the study is to establish a relationship between the administered activity of the radioiodine and absorbed dose in the tumor sites.

DETAILED DESCRIPTION:
Study Design - the assessment of patients with multiple tumour sites with metastatic thyroid cancer to correlate the administered activity to absorbed dose. Patients will receive the standard therapy dose of 5.5 GBq as per the hospital policy and there will be no change for the protocol purpose.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* histological confirmation of the differentiated thyroid carcinoma available
* WHO performance score 0-2
* metastatic sites lung and/or bone and/or nodal (radiologically measurable disease > 1 cm)
* life expectancy > 6 months
* patient has undergone total/near total thyroidectomy
* no past history of sensitivity/reaction to 1311

Exclusion Criteria:

* non iodine concentrating tumours
* received chemotherapy or radiotherapy in 6 weeks
* pregnant or breast feeding patients
* iodine contrast injection in last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-01 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is to correlate the predicted dose from the tracer study with the actual absorbed dose measure on the therapeutic scan

SECONDARY OUTCOMES:
The secondary outcomes will be to assess the response at 6 months post therapy in each patient

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kate Newbold, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, Sutton, United Kingdom